CLINICAL TRIAL: NCT01178879
Title: Effectiveness of Nurse Lead Telehealth Consultations in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Randomised Trial of Telehealth Consultations for Nursing Care of Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Sygekassernes Helsefond (Other); Danish Nurses Organisation (Other)
Responsible Party: Principal Investigator, Birte Oestergaard, Associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNRS-20100030-2
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: COPD
Keywords: Telehealth; nurse consultation; outpatient clinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telehealth consultation (Experimental): Telehealth nurse consultation plus treatment as usual
  Interventions: Behavioral: Telehealth consultation
- Conventional (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Telehealth consultation — The consultations are structured as outpatient sessions immediately after discharge. The content of the education deals with the regular treatment, prevention of exacerbation and how to live with the illness. The aim of the counseling is to increase the patient's empowerment and competence to take action. The patients have the consultations for 7 days followed by a telephone call. Each session is organized and individualised according to the patient's wishes and needs for education and counselling.
  The equipment consists of a computer with web camera, microphone and measurement equipment. A button to contact to the nurse at the hospital, an alarm button and a volume button. The results are transferred to the hospital by a secure internet line.
  Other Names: Telehealth nurse consultation
  Arms: Telehealth consultation

SUMMARY:
The purpose of this study is to determine whether telehealth nursing consultations of chronic obstructive pulmonary disease (COPD) patients are superior to hospital readmissions.

DETAILED DESCRIPTION:
COPD is among the most common reasons for illness and fatality in adults worldwide, and it is expected that this trend will escalate radically by 2020 (1). Approximately 29% of patients admitted to Hospital with exacerbation will be readmitted within the first month (2), and after one year 46% of patients will have been readmitted on one or more occasions due to exacerbation (3).

Therefore, trials have been carried out using different forms of digitally supported distance health interventions (telehealth nurse consultations) (4) of patients with COPD with a view to reducing the number of readmissions in a reliable way, measured in relation to mortality. Thus in these trials there are a certain indication that use of telehealth nurse consultations of patients with COPD is a treatment initiative that reliably can reduce the number of COPD patients readmitted with exacerbation.

The number of randomized telehealth studies are however few (4;5), and there is a lack of documentation of the effect of telehealth monitoring.

Therefore, a large randomized telehealth study with a clear set up was necessary.

This study is a randomized multicenter trial that will take place at the acute admissions department and lung department at Odense University Hospital,Denmark

We hypothesized that in a period of 26 weeks:

1. The total number of readmissions can be reduced with 14%
2. The time to the first readmission will be prolonged
3. The number of readmissions with exacerbation can be reduced after telehealth consultations as a supplement to the conventional treatment compared with conventional treatment
4. The total number of readmission days can be reduced after telehealth consultations as a supplement to the conventional treatment compared with conventional treatment
5. The total number of readmission days with exacerbation can be reduced after telehealth consultations as a supplement to the conventional treatment compared with conventional treatment
6. The mortality rate will remain unchanged after the telehealth consultations as a supplement to the conventional treatment compared with conventional treatment

ELIGIBILITY:
Inclusion criteria:

* Chronic obstructive pulmonary disease (COPD) verified by spirometry.
* Exacerbation in COPD, defined as increased need for medicine, and increased dyspnea or increased expectorate or increased coughing.
* > or 40 years old
* Living on Funen and islands
* Signed informed consent.

Exclusion criteria:

* Not able to communicate via telephone and/or computer screen
* Previously received "The COPD suitcase", or participated in this protocol
* Systolic BT is <100 mm Hg
* Saturation < 90
* Thorax x-ray shows signs of malignant changes or lobar pneumonia
* Diagnosed with cancer or recurrence of cancer within the last five years
* Admitted with septic shock, acute myocardial infarction or other serious medical condition (for example renal disease)
* Diagnosed with heart failure (EF < 30%)
* Refused to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The number of readmissions | at 26 weeks after discharge

SECONDARY OUTCOMES:
The mortality rate | at 26 weeks weeks after discharge
The duration to the first readmission | at 26 weeks after discharge
The number of hospital readmissions with exacerbation | at 26 weeks after discharge
The number of days readmitted | days 26 weeks after discharge
The number of days readmitted with exacerbation | days 26 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dichmann Sorknaes, PhD student, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Murray CJ, Lopez AD. Alternative projections of mortality and disability by cause 1990-2020: Global Burden of Disease Study. Lancet. 1997 May 24;349(9064):1498-504. doi: 10.1016/S0140-6736(96)07492-2. PMID 9167458
- [Background] (2) Sundhedsstyrelsen. Genindlæggelser af ældre i Danmark 2008 - Nye tal fra Sundhedsstyrelsen. 1060. Ref Type: Internet Communication.
- [Background] Eriksen N, Hansen EF, Munch EP, Rasmussen FV, Vestbo J. [Chronic obstructive pulmonary disease. Admission, course and prognosis]. Ugeskr Laeger. 2003 Sep 8;165(37):3499-502. Danish. PMID 14531348
- [Background] Casas A, Troosters T, Garcia-Aymerich J, Roca J, Hernandez C, Alonso A, del Pozo F, de Toledo P, Anto JM, Rodriguez-Roisin R, Decramer M; members of the CHRONIC Project. Integrated care prevents hospitalisations for exacerbations in COPD patients. Eur Respir J. 2006 Jul;28(1):123-30. doi: 10.1183/09031936.06.00063205. Epub 2006 Apr 12. PMID 16611656
- [Background] Finkelstein SM, Speedie SM, Potthoff S. Home telehealth improves clinical outcomes at lower cost for home healthcare. Telemed J E Health. 2006 Apr;12(2):128-36. doi: 10.1089/tmj.2006.12.128. PMID 16620167